CLINICAL TRIAL: NCT07359248
Title: Study on the Effectiveness of Preventive Treatment With Venlafaxine for Frequent Episodic Tension-type Headache
Brief Title: Desvenlafaxine for Preventive Treatment of Frequent Episodic Tension-type Headache
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wensheng Qu, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20251111TTH
Record Dates: First submitted 2025-11-26; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: Tension Type Headache
MeSH Terms: conditions — Tension-Type Headache | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desvenlafaxine (Experimental): Participants in this arm will receive oral Desvenlafaxine at a fixed dose of 50 mg once daily for 12 weeks.
  Interventions: Drug: Desvenlafaxine
- placebo (Placebo Comparator): Participants in this arm will receive an identical-appearing placebo tablet administered orally once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desvenlafaxine — Desvenlafaxine
  Arms: Desvenlafaxine
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
To evaluate whether Desvenlafaxine can reduce the frequency and severity of TTH attacks in patients.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled trial aims to assess the efficacy of Desvenlafaxine (a serotonin-norepinephrine reuptake inhibitor) in reducing the frequency and severity of tension-type headache (TTH) attacks in adult patients with episodic TTH.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18-65 years
2. Meeting the diagnostic criteria for tension-type headache (TTH) according to ICHD-3; with ≥6 but <15 attack days per month in the past 3 months and MIDAS score >21; onset of TTH before age 50, with a history exceeding 1 year
3. Informed consent obtained from the patient

Exclusion Criteria:

1. History of allergy to Desvenlafaxine, or use of Desvenlafaxine within 4 weeks prior to the start of the treatment period; currently taking or requiring concomitant administration of drugs contraindicated in the package insert, such as monoamine oxidase inhibitors (MAOIs);
2. Diagnosable with chronic tension-type headache or medication overuse headache;
3. Comorbid with other types of headaches, such as trigeminal autonomic cephalalgias, migraine attacks >1 time/month within 3 months, or secondary headaches (e.g., those caused by intracranial infections, craniocerebral trauma, cerebrovascular diseases);
4. Severe psychiatric disorders such as schizophrenia, moderate to severe anxiety-depression (Hamilton scale ≥12 points); poorly controlled epilepsy, cognitive impairments, and other chronic pain conditions; serious organic diseases that pose significant health risks, including uncontrolled hypertension, cardiac disease, hepatic dysfunction, renal insufficiency, infections; any medical condition or prior surgery likely to affect the absorption, metabolism, or excretion of the study drug;
5. Concomitant use of venlafaxine analogues such as serotonin-norepinephrine reuptake inhibitors (SNRIs); unstable use of other preventive medications for TTH, including amitriptyline, mirtazapine (≤3 months); discontinuation of currently reported effective prophylactic drugs or overused analgesics for ≥3 months may allow re-enrollment;
6. Alcohol dependence or substance abuse;
7. Inability to comprehend the study protocol due to low education level, impaired verbal/language function, visual or auditory deficits; failure to accurately complete research materials like headache diaries or cooperate with scale assessments;
8. Women who are planning pregnancy, pregnant, breastfeeding, or not using contraception;
9. Participation in other interventional clinical studies that may influence outcome evaluations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Days with tension-type headache (TTH) during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12) | During the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
  Days with tension-type headache (TTH) during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)

SECONDARY OUTCOMES:
Total headache index AUC (area under the curve) during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12) | during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
  Total headache index AUC (area under the curve) during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
Headache severity (VAS 0-10) and duration (hours per day) during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12) | during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
  Headache severity (VAS 0-10) and duration (hours per day) during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
Acute analgesic consumption: number of days and dosage | during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
  Acute analgesic consumption: number of days and dosage
Treatment effectiveness criterion: reduction in headache days by ≥50% during the third 4-week intervention period compared to the screening period | during the third 4-week intervention period
  Treatment effectiveness criterion: reduction in headache days by ≥50% during the third 4-week intervention period compared to the screening period
Safety assessment and tolerability evaluation | During the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
  Safety and tolerability will be evaluated by: Continuous recording of treatment-emergent adverse events (TEAEs, graded by CTCAE v5.0) throughout the study.
Change in headache impact on daily life as assessed by the 6-item Headache Impact Test (HIT-6) total score | During the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
  The HIT-6 questionnaire measures the adverse impact of headache on daily functioning in six domains (pain, social functioning, role functioning, vitality, cognitive functioning, psychological distress).

CONTACTS AND LOCATIONS:
Overall Officials: Wensheng Qu, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
No immediate plans exist for IPD sharing, but controlled access may be considered post-study completion